CLINICAL TRIAL: NCT04583358
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Multicenter, Phase 2a Study of the Efficacy and Safety of Oral AMT-101 in Subjects With Moderate to Severe Ulcerative Colitis (LOMBARD)
Brief Title: Study of the Efficacy and Safety of AMT-101 in Subjects With Ulcerative Colitis (LOMBARD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Applied Molecular Transport (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMT-101-202
Record Dates: First submitted 2020-09-16; First posted 2020-10-12 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMT-101 (Active Comparator): AMT-101 Tablet
  Interventions: Drug: AMT-101 (oral)
- Placebo (Placebo Comparator): Placebo Tablet
  Interventions: Other: Placebo (oral)

INTERVENTIONS:
Drug: AMT-101 (oral) — AMT 101 is orally administered biological therapeutic taken once daily
  Arms: AMT-101
Other: Placebo (oral) — Orally administered placebo comparator taken once daily
  Arms: Placebo

SUMMARY:
Randomized, Placebo-controlled, Double-blind, Parallel-group, Multicenter, Phase 2a Study of the Efficacy and Safety of Oral AMT-101 in Subjects with Moderate to Severe Ulcerative Colitis.

DETAILED DESCRIPTION:
This is a Randomized, Placebo-controlled, Double-blind, Parallel-group, Multicenter, Phase 2a Study to evaluate the Efficacy and Safety of Oral AMT-101 in Subjects with Moderate to Severe Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 75 years, inclusive.
* Diagnosis of moderate to severe UC.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and at the randomization visit.
* Able to participate fully in all aspects of this clinical trial.
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Known gastrologic, or systemic condition that may compromise severity or diagnosis of disease.
* History or current evidence of colonic or abdominal abnormalities.
* Prohibited therapies or procedures before the screening period as specified per protocol.
* A concurrent clinically significant, serious, unstable, or uncontrolled underlying cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, might confound the study results, pose additional risk to the subject, or interfere with the subject's ability to participate fully in the study.
* Pregnant or lactating females.
* Current or recent history of alcohol dependence, illicit drug use, mental or legal incapacitation, or a history of clinically significant psychiatric disorders that, in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures.
* Unable to attend study visits or comply with procedures.
* Previous exposure to AMT-101 or similar and known hypersensitivity to AMT-101 or its excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mayo Score | 12 weeks

SECONDARY OUTCOMES:
Endoscopic Remission Rate | 12 weeks
Mucosal Healing Rate | 12 weeks
Histologic Remission Rate | 12 weeks
Clinical Remission Rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (59):
- United States (15):
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - AdventHealth - Florida Hospital, Orlando, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Gwinnett Research Institute, LLC, Buford, Georgia
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Carolina Research, Greenville, North Carolina
  - Gastro One, Germantown, Tennessee
  - GIA Clinical Trials, LLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Caprock Gastro Research, Lubbock, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Washington Gastroenterology, Bellevue, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
- Vitebsk Regional Clinical Hospital, Vitebsk, Vitebsk Oblast, Belarus
- Bulgaria (2):
  - MHAT Blagoevgrad AD, Blagoevgrad
  - MHAT Lyulin EAD, Sofia
- Canada (3):
  - GI Research Institute, Vancouver, British Columbia
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Toronto Digestive Disease Associates Specialty Research, Vaughan, Ontario
- CHU Saint-Etienne - Hospital Nord Gastroenteroloy, Saint-Priest-en-Jarez, France
- Arensia Exploratory Medicine GmbH, Tbilisi, Georgia
- Germany (4):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Jena Klinik fuer Innere Medizin IV, Jena, Thuringia
  - University Hospital Schleswig-Holstein, Kiel
  - Staedtisches Klinikum Lueneburg, Lüneburg
- Hungary (5):
  - Mohacsi Korhaz, Mohács, Baranya
  - Szegedi Tudomanyegyetem, Szeged, Csongrád megye
  - Javorszky Odon Korhaz, Gasztroenterologiai Osztaly, Vác, Pest County
  - Clinexpert Kft., Budapest
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest
- Clinical Republican Hospital "Timofei Mosneaga", ARENSIA E.M., Chisinau, Municipality of Chisinau, Moldova
- Poland (12):
  - Centrum Medyczne CLW-MED, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Kopon, Zmudziski I Wspolnicy Sp.j., Torun, Kuyavian-Pomeranian Voivodeship
  - Vistamed & Vertigo Sp. z o.o, Wroclaw, Lower Silesian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovia
  - Nzoz Vivamed, Warsaw, Masovia
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Centrum Medyczne LUKAMED Joanna Luka-Wendrowska, Chojnice, Pomeranian
  - Indywidualna Praktyka Lekarska Maciej Zymła, Knurów, Silesian
  - Vitamed Gałaj i Cichomski S.J., Bydgoszcz
  - Centrum Medyczne Medyk, Rzeszów
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska S.J., Ksawerów, Łódź Voivodeship
  - Nowe Zdrowie CK Kieltucki I Wspólnicy sp.j., Staszów, Świętokrzyskie Voivodeship
- Russia (2):
  - Novosibirsk GastroCenter LLC, Novosibirsk, Novosibirsk Oblast
  - Medical Diagnostics Center, LLC, Yaroslavl, Yaroslavl Oblast
- Clarunis Bauchzentrum, Basel, Switzerland
- Ukraine (10):
  - Regional Hospital of War Veterans, Kharkiv
  - Medical and Diagnostic Centre of Private Enterprise of Private Manufacturing Company "Acinus", Kropyvnytskyi
  - Medical center limited liability Harmoniya Krasy, Kyiv
  - Medical Center Ok!Clinic+ International Institute, Kyiv
  - CI of Kyiv RC Regional Clinical Hospital No 2, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Uzhgorod National University, Uzhhorod
  - Vinnytsya City Clinical Hospital No 1, Vinnytsia
  - Medical Center of Limited Liability Co, Zaporizhzhia
  - Limited Liability Company Medibor, Zhytomyr
- Barnsley Hospital NHS Foundation Trust, Barnsley, Yorkshire, United Kingdom